CLINICAL TRIAL: NCT02192606
Title: Does 3D Laparoscopy Improve Vaginal Cuff Suture Time? A Randomized Controlled Trial Comparing 3D Laparoscopy Versus Standard Laparoscopy
Brief Title: Does 3D Laparoscopy Improve Vaginal Cuff Suture Time?
Acronym: 3DRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jon I. Einarsson, Division Chair, Minimally Invasive Gynecology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3DRCT
Record Dates: First submitted 2013-11-05; First posted 2014-07-17 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Uterine Fibroids; Abnormal Uterine Bleeding; Pelvic Pain; Adenomyosis
Keywords: Laparoscopy; 3D Visual System; Total Hysterectomy
MeSH Terms: conditions — Leiomyoma; Metrorrhagia; Pelvic Pain; Adenomyosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2D Laparoscopy (Active Comparator): The standard 2D Laparoscopy System to be used at time of the total laparoscopic hysterectomy
  Interventions: Device: 2D Laparoscopy
- 3D laparoscopy (Active Comparator): The Storz 3D Laparoscopy System is the intervention we are studying at the time of the total laparoscopic hysterectomy.
  Interventions: Device: Storz 3D Laparoscopy System

INTERVENTIONS:
Device: Storz 3D Laparoscopy System — The Storz 3D Laparoscopy System is a new device that allows for laparoscopic surgeons to utilize 3D imaging during surgery with a fraction of the cost of the da Vinci Surgical System, a three-dimensional visual system.
  Arms: 3D laparoscopy
Device: 2D Laparoscopy — The standard 2D Laparoscopy System to be used at time of the total laparoscopic hysterectomy.
  Arms: 2D Laparoscopy

SUMMARY:
The objective aim is to evaluate whether the use of 3D laparoscopy facilitates the vaginal cuff closure of the vaginal cuff during a total laparoscopic hysterectomy among novice laparoscopists (PGY 2-4, Fellow). This is a randomized single blinded controlled trial comparing the difference in 2D vs. 3D in regards to vaginal cuff closure time stratified by residents and fellows. Patients will undergo a total laparoscopic hysterectomy and will be randomized to either 2D versus 3D.

DETAILED DESCRIPTION:
This is a randomized single blinded controlled trial investigating 3D laparoscopy in the clinical setting. Based on previous studies indicating 3D laparoscopy has improved skills of novice surgeons in the simulation lab, there has been no reports to date investigating the role of 3D laparoscopy in the operating room. Our study will evaluate the facility of 3D laparoscopy in the novice surgeon, mainly residents and fellow. Patients who present for a scheduled total laparoscopic hysterectomy will be randomized to either the standard 2D laparoscopy system or 3D laparoscopy system. Stratifying residents versus fellow, we will compare the time to close the vaginal cuff comparing both systems.

ELIGIBILITY:
Inclusion Criteria:

* Women with benign conditions such as uterine fibroids, menorrhagia, adenomyosis, pelvic pain, abnormal uterine bleeding

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Einarsson, MD, PhD, MPH, Principal Investigator — Brigham and Women's Hospital; Sarah L Cohen, MD, MPH, Study Director — Brigham and Women's Hospital
Locations (2):
- Brigham & Women's Hospital, Boston, Massachusetts, United States
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhayani SB, Andriole GL. Three-Dimensional (3D) Vision: Does It Improve Laparoscopic Skills? An Assessment of a 3D Head-Mounted Visualization System. Rev Urol. 2005 Fall;7(4):211-4. PMID 16985832
- [Background] Tanagho YS, Andriole GL, Paradis AG, Madison KM, Sandhu GS, Varela JE, Benway BM. 2D versus 3D visualization: impact on laparoscopic proficiency using the fundamentals of laparoscopic surgery skill set. J Laparoendosc Adv Surg Tech A. 2012 Nov;22(9):865-70. doi: 10.1089/lap.2012.0220. Epub 2012 Oct 16. PMID 23072406
- [Background] Einarsson JI, Wang KC, Cohen SL, Sandberg EM, Vree FEM, Jonsdottir GM, Gobern J, Brown DN. A Randomized Controlled Trial of Barbed versus Traditional Suture for Vaginal Cuff Closure at Time of Total Laparoscopic Hysterectomy: Preliminary Results. Abstracts/ Journal of Minimally Invasive Gynecology. 19 (2012); S36-70.
- [Derived] Ajao MO, Larsen CR, Manoucheri E, Goggins ER, Rask MT, Cox MKB, Mushinski A, Gu X, Cohen SL, Rudnicki M, Einarsson JI. Two-dimensional (2D) versus three-dimensional (3D) laparoscopy for vaginal cuff closure by surgeons-in-training: a randomized controlled trial. Surg Endosc. 2020 Mar;34(3):1237-1243. doi: 10.1007/s00464-019-06886-9. Epub 2019 Jun 6. PMID 31172324

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2D Laparoscopy | 3D Laparoscopy
Started | 29 | 28
Completed | 27 | 24
Not Completed | 2 | 4
Not completed — surgery type was changed | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — 3D equipment rep unable to join | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2D Laparoscopy | 3D Laparoscopy | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (5.2) | 43.9 (8.2) | 42.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
  Denmark | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Cuff Closure Times
Description: The primary endpoint is the vaginal cuff closure time at the time of a total laparoscopic hysterectomy. As the 2D laparoscopy system is standard during laparoscopic cases, our objective is to assess if there is a difference in vaginal cuff closure time when a 3D laparoscopy system is used instead. At time of the surgery, that patient will be randomized to either system. A resident or fellow will close the vaginal cuff and time to close the vaginal cuff will be recorded.
Time Frame: Start of vaginal cuff closure to end of vaginal cuff closure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 2D Laparoscopy | 3D Laparoscopy
Number analyzed (Participants) | 29 | 28
minutes | 10.17 (5.98) | 12.54 (6.99)

2. Secondary Outcome: Estimated Blood Loss at the Time of Total Laparoscopic Hysterectomy
Description: The secondary endpoint is the surgeon estimated blood loss at the time of a total laparoscopic hysterectomy.
Time Frame: Time of Procedure End
Measure: Mean (Standard Deviation); unit: millileters
Arm/Group | 2D Laparoscopy | 3D Laparoscopy
Number analyzed (Participants) | 29 | 28
millileters | 55.74 (39.36) | 60.83 (62.32)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the day of surgery to 8 weeks following the operation.
Arm/Group | 2D Laparoscopy | 3D Laparoscopy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 3/29 | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2D Laparoscopy (N=29) | 3D Laparoscopy (N=28)
ER visit (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject presented to ER 5 days after discharge concerned about blood clot in hand where IV had been. Seen and prescribed warm compresses and discharged.
Reoperation for vaginal cuff dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1) — Subject presented to ER 18 days after surgery with abdominal pain. Rxed with dilaudid; required re-operation for cuff dehiscence.
Iritation around abdominal surgical incision site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject experienced some postoperative red/itching around incision sites - near smaller incisions like a rash; advised oral antihistamines and topical hydrocortisone for presumed dermabond reaction. Improved with treatment.
Incision cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Subject was treated with antibiotics for postoperative incision cellulitis.
Yeast infection (Infections and infestations) | 1 (1) | 0 (0) — Subjected was treated with diflucan for postoperative yeast infection.
Intraoperative complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Intraoperative cystotomy (bladder injury), repaired laparoscopically. Normal recovery.
Urinary retention (General disorders) | 1 (1) | 0 (0) — Subject had postoperative urinary retention with transient Foley catheter needed but returned to normal by post-operative follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No